CLINICAL TRIAL: NCT03017274
Title: Abdominal Ultrasound Examination in Patients Affected With Non-celiac Wheat Sensitivity
Brief Title: Abdominal Ultrasound Examination in Non-celiac Wheat Sensitivity
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM20
Record Dates: First submitted 2016-12-30; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac wheat sensitivity; celiac disease; abdominal ultrasonography;
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NCWS patients: Fifty consecutive adult patients with an IBS-like clinical presentation, according to Rome III criteria, and a definitive diagnosis of NCWS. The patients was recruited between January 2015 and November 2016 at 2 centers: the Department of Internal Medicine at the University Hospital of Palermo, Italy, and the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy. All subjects undergone abdominal ultrasonography at the Outpatient of Ultrasonography of the Department of Internal Medicine at the University Hospital of Palermo, Italy.
  Interventions: Other: Abdominal ultrasound examination
- CD control patients: To compare the abdominal ultrasonographic features of NCWS patients, a control group of CD patients was randomly chosen by a computer-generated method from subjects diagnosed during the same period and age- and sex-matched with the NCWS patients. All subjects undergone abdominal ultrasonography at the Outpatient of Ultrasonography of the Department of Internal Medicine at the University Hospital of Palermo, Italy.
  Interventions: Other: Abdominal ultrasound examination

INTERVENTIONS:
Other: Abdominal ultrasound examination — All subjects undergone abdominal ultrasonography at the Outpatient of Ultrasonography of the Department of Internal Medicine at the University Hospital of Palermo, Italy.

SUMMARY:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays no data are available on the abdominal ultrasonographic features of NCWS patients. Therefore, the aim of the present study is to evaluate the abdominal ultrasonographic features of NCWS patients in comparison with patients affected with celiac disease.

DETAILED DESCRIPTION:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). The researchers have just demonstrated in patients affected with seronegative celiac disease that the presence of dilated bowel loops and a thickened small bowel wall had a sensitivity of 83% and a negative predictive value of 95% in CD diagnosis. Considering the presence of one of these two signs, abdominal US sensitivity increased to 92% and negative predictive value to 98%. Nowadays no data are available on the abdominal ultrasonographic features of NCWS patients. Therefore, the aim of the present study is to evaluate the abdominal ultrasonographic features of NCWS patients in comparison with patients affected with celiac disease.

ELIGIBILITY:
Inclusion Criteria:

To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* absence of intestinal villous atrophy
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection)
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.

To diagnose CD the standard criteria will be adopted. All the patients will meet the following criteria:

* positive serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* presence of intestinal villous atrophy.

Exclusion Criteria:

NCWS diagnosis excluded patients with:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other previously diagnosed gastrointestinal disorders
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included consecutive adult patients with IBS-like clinical presentation, according to Rome III criteria, and a definitive diagnosis of NCWS, referred at the Department of Internal Medicine at the University Hospital of Palermo, Italy, and at the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy, between January 2015 and November 2016, and sex- and age-matched subjects with CD, enrolled at the same centers, as controls patients. All subjects undergone abdominal ultrasonography at the Outpatient of Ultrasonography of the Department of Internal Medicine at the University Hospital of Palermo, Italy.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Abdominal ultrasonographic features of NCWS and CD patients | from January 2015 to November 2016
  Evaluation of abdominal ultrasonographic differences between NCWS and CD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Soresi M, Pirrone G, Giannitrapani L, Iacono G, Di Prima L, La Spada E, Di Fede G, Ambrosiano G, Montalto G, Carroccio A. A key role for abdominal ultrasound examination in "difficult" diagnoses of celiac disease. Ultraschall Med. 2011 Jan;32 Suppl 1:S53-61. doi: 10.1055/s-0028-1110009. Epub 2010 Mar 16. PMID 20235005
- [Derived] Soresi M, Mansueto P, Terranova A, D'Alcamo A, La Blasca F, Cavataio F, Iacobucci R, Carroccio A. Abdominal Ultrasound Does Not Reveal Significant Alterations in Patients With Nonceliac Wheat Sensitivity. J Clin Gastroenterol. 2019 Jan;53(1):e31-e36. doi: 10.1097/MCG.0000000000000969. PMID 29206754